CLINICAL TRIAL: NCT01466725
Title: A Phase 2, Pilot, Multicenter, Randomized, Placebo-Controlled Sequential, Ascending Dose Study to Characterize the Safety, Tolerability, Pharmacokinetic and Pharmacodynamic Activity of CC-930 in Subjects With Recalcitrant Discoid Lupus Erythematosus (DLE)
Brief Title: A Research Study to Assess if CC-930 is Safe in Treating Subjects With Discoid Lupus Erythematosus
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The benefit/risk profile does not support continuation of this study.
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CC-930-DLE-002
Record Dates: First submitted 2011-11-04; First posted 2011-11-08 (Estimated); Last update posted 2019-11-19 (Actual); Status verified 2019-11

CONDITIONS: Discoid Lupus
Keywords: Lupus; Discoid Lupus; DLE; Cutaneous Lupus
MeSH Terms: conditions — Lupus Erythematosus, Discoid | interventions — 4-(9-(tetrahydrofuran-3-yl))-8-(2,4,6-trifluorophenylamino)-9H-purin-2-ylaminocyclohexan-1-ol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Cohort 1 (Experimental): 25 mg daily for 4 weeks (8 active/2 control)
  Interventions: Drug: CC-930; Drug: Placebo
- Cohort 2 (Experimental): 50 mg once daily for 4 weeks (8 active/2 control)
  Interventions: Drug: CC-930; Drug: Placebo
- Cohort 3 (Experimental): 100 mg daily for 6 weeks (8 active/2 control)
  Interventions: Drug: CC-930; Drug: Placebo
- Cohort 4 (Experimental): 100 mg twice daily for 6 weeks (8 active/2 control)
  Interventions: Drug: CC-930; Drug: Placebo

INTERVENTIONS:
Drug: CC-930
Drug: Placebo — Placebo

SUMMARY:
The purpose of the study is to assess if CC-930 is safe and tolerable in treating subjects with Discoid Lupus Erythematosus. Pharmacokinetic and pharmacodynamics will also be evaluated.

DETAILED DESCRIPTION:
Enrollment will occur in sequential, ascending, dose-sequence design, where a higher CC-930 dose level and longer duration of dosing (cohort) will not be initiated until supportive safety profile is demonstrated in the preceding cohort. There will be 4 cohorts as described here;

Cohort 1: 25 mg once daily for 4 weeks Cohort 2: 50 mg once daily for 4 weeks Cohort 3: 100 mg once daily for 6 weeks Cohort 4: 100 mg twice daily for 6 weeks

ELIGIBILITY:
Inclusion Criteria:

1. Male or female with clinical diagnosis of Discoid Lupus Erythematosus (DLE) aged 18 to 64 years
2. Good health as assessed by Investigator
3. DLE for at least 16 weeks prior to screening and consistent histological findings.
4. Considered a candidate for systemic therapy. May be naïve to systemic therapy or experiencing incomplete or refractory disease on systemic therapy.
5. Cutaneous Lupus Area and Severity Index (CLASI) activity score of at least 10, as determined by investigator.
6. Subjects using hydroxychloroquine, chloroquine, or quinacrine must have documented ophthalmologic exam within 24 weeks of baseline visit.
7. Must meet laboratory criteria for white blood cells, absolute neutrophils, platelets, serum creatinine, aspartate aminotransferase (AST), alanine aminotransferase (ALT), bilirubin and hemoglobin.
8. Subjects, male and female, must agree to strict pregnancy prevention and testing requirements.

Exclusion Criteria:

1. Significant illnesses as determined by physician.
2. History of significant cardiac conditions or interventions within prior 6 months including abnormal electrocardiogram (ECG) findings.
3. Systolic blood pressure < 95 or > 150 mm Hg
4. Diastolic blood pressure > 90 mm Hg.
5. Pregnancy or breast feeding.
6. Other dermatological conditions that would interfere with CLASI Activity Score assessments.
7. History of or active; malignancy, human immunodeficiency virus (HIV), tuberculosis infection, other mycobacterial infection, congenital or acquired immunodeficiency, Hepatitis B and C.
8. Clinically significant abnormality on chest X-ray.
9. Participation in multiple CC-930 cohorts.
10. History of thrombolytic event.
11. Positive tests for lupus anticoagulant, anti-cardiolipin antibodies, antibodies to beta-2 glycoprotein 1 or phosphatidylserine at screening.
12. Positive antineutrophilic cytoplasmic antibody (ANCA) at screening.
13. Diagnosis of SLE.
14. Presence or history of medically significant Systemic Lupus Erythematosis (SLE) or Lupus Erythematosis (LE) comorbidities.
15. History of seizures, chorea or psychosis.
16. Presence or history of persistent proteinuria or urinary cellular casts.
17. Prohibited prior or concomitant medications.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2011-11-01 (Actual); Primary Completion 2012-07-30 (Actual); Study Completion 2012-07-30 (Actual)

PRIMARY OUTCOMES:
Number of subjects with adverse events | 4 to 6 weeks

SECONDARY OUTCOMES:
To describe the pharmacokinetics of CC-930 in subjects with recalcitrant DLE. | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: William Smith, MD, Study Director — Celgene
Locations (19):
- United States (19):
  - UAB Dermatology, Birmingham, Alabama
  - The Regents of the University of California, Irvine, California
  - Medical Faculty Associates, Washington D.C., District of Columbia
  - Advanced Pharma, CR, LLC, Miami, Florida
  - University of Miami - Department of Dermatology, Miami, Florida
  - Rush Medical Center, Chicago, Illinois
  - North Shore University Health System, Skokie, Illinois
  - SIU School of Medicine, Springfield, Illinois
  - Tulane University School of Medicine, New Orleans, Louisiana
  - John Hopkins University, Baltimore, Maryland
  - Boston Cancer Center, Boston, Massachusetts
  - University of Minnesota-Department of Dermatology, Minneapolis, Minnesota
  - University of Rochester Medical Center, Rochester, New York
  - Ohio State Univ Medical Center, Division of Dermatology, Columbus, Ohio
  - Rhode Island Hospital University Dermatology, Inc., Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - Dermatology and Research, Dallas, Texas
  - University of Texas Dermatology, Houston, Texas
  - Sun Research Institute, San Antonio, Texas